CLINICAL TRIAL: NCT04280029
Title: SELUTION SLR™ 014 ISR: A Prospective Randomized Single Blind Multicenter Study to Assess the Safety and Effectiveness of the SELUTION SLR™ 014 Drug Eluting Balloon in the Treatment of Subjects With In-stent Restenosis
Brief Title: SELUTION SLR™ 014 In-stent Restenosis
Acronym: SELUTION4ISR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEL-003-2019
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Coronary Restenosis
Keywords: In-stent restenosis; Drug Eluting Balloon; Coronary
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- SELUTION SLR 014 DEB (Experimental): The SELUTION Sustained Limus Release (SLR)™ 014 drug-eluting balloon (DEB) catheter is a combination product consisting of a standard percutaneous transluminal angioplasty (PTA) balloon catheter coated with a drug (Sirolimus).
  Interventions: Device: SELUTION SLR 014 DEB
- Standard Of Care (Active Comparator): POBA or FDA-approved commercially available -limus eluting DES
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: SELUTION SLR 014 DEB — The SELUTION Sustained Limus Release (SLR)™ 014 drug-eluting balloon (DEB) catheter is a combination product consisting of a standard percutaneous transluminal angioplasty (PTA) balloon catheter coated with a drug (Sirolimus).
  Arms: SELUTION SLR 014 DEB
Device: Standard of Care — POBA or FDA-approved commercially available -limus eluting DES
  Arms: Standard Of Care

SUMMARY:
Prospective, multi-center, randomized, single blind, controlled, noninferiority clinical trial.

Subjects with previous bare-metal stent (BMS) or DES and qualifying evidence for ISR will be screened per the protocol inclusion and exclusion criteria. Eligible subjects will be randomized 1:1 to treatment with either the SELUTION SLR 014 DEB or SOC to include contemporary DES (zotarolimus-eluting stents [ZES] and everolimus-eluting stents [EES] only) or BA. A maximum of 20% of patients randomized to SOC will be treated with BA.

The primary endpoint will be Target Lesion Failure (TLF) at 12-months in the SOC group vs. the SELUTION SLR 014 DEB in all patients.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized, single blind, controlled, noninferiority clinical trial will enroll up to 418 randomized subjects (including up to 60 subjects in an angiographic and optical coherence tomography [OCT] sub-study) at up to 80 sites in the United States (US), Canada, Brazil, and Europe (EU). A minimum of 50% of the subjects will be enrolled in the US.

Subjects with previous bare-metal stent (BMS) or DES and qualifying evidence for ISR will be screened per the protocol inclusion and exclusion criteria. Eligible subjects will be randomized 1:1 to treatment with either the SELUTION SLR 014 DEB or SOC to include contemporary DES (zotarolimus-eluting stents [ZES] and everolimus-eluting stents [EES] only) or BA. A maximum of 20% of patients randomized to SOC will be treated with BA.

The primary endpoint will be Target Lesion Failure (TLF) at 12-months in the SOC group vs. the SELUTION SLR 014 DEB group.

A subset of up to 60 subjects will be enrolled in the angiographic and OCT sub-study and undergo planned angiographic and OCT follow-up within 30 days after completion of the 12-month primary endpoint clinical follow-up/assessment.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject age is ≥ 18 years or minimum legal age as required by local regulations.
2. Female subjects of childbearing potential have a negative pregnancy test ≤ 7 days before the procedure.
3. Subject presents with chronic coronary syndrome (CCS) (manifest as documented angina or positive functional testing), unstable angina or stabilized non-ST-elevation myocardial infarction (NSTEMI) (biomarkers stabilized or down trending) with an indication for percutaneous coronary intervention (PCI) and planned intervention.
4. Subject is eligible for dual antiplatelet therapy (DAPT) treatment with aspirin plus either Clopidogrel, Prasugrel, or Ticagrelor. Note: Subjects who require continued oral anticoagulant therapy my omit aspirin at discretion of investigator.
5. Life expectancy >1 year in opinion of investigator.
6. Subject is willing and able to provide informed consent and comply with study procedures and required follow-up evaluations.

Angiographic Inclusion Criteria

1. Target lesion is within a native coronary artery or major branch.
2. Target lesion is within a previously placed BMS or DES and does not extend further than 5 mm beyond either the proximal or distal edge of the stent.
3. Up to two (2) non-target lesions in non-target vessels may be treated, but successful PCI of the non-target lesions must be completed before treatment of the target lesion. Successful treatment is defined as no greater than 30% residual stenosis by visual estimate, no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C, and Thrombolysis in Myocardial Infarction (TIMI) grade flow in the non-target lesion > 2.
4. Target lesion is ≤ 26 mm in length.
5. Target lesion has diameter stenosis of > 50% and ≤ 99% by visual estimate.
6. Reference vessel diameter (RVD) is ≥ 2.00 mm and ≤ 4.50 mm.
7. Target lesion must be successfully pre-dilated/pre-treated. Note: Successful pre-dilation/pre-treatment is defined as dilation or pre-treatment that achieves stent expansion of approximately 80% of the distal RVD (at the discretion of the investigator) based on intravascular ultrasound (IVUS)/optical coherence tomography (OCT) and no greater than 30% residual stenosis by visual estimate and no dissection greater than NHLBI type C. TIMI grade flow in the target lesion must be > 2. Note: Atherectomy and cutting balloon are permitted for pre-treatment.

Clinical Exclusion Criteria:

1. Known hypersensitivity or allergy to Sirolimus or other pharmacologic agents required for the procedure.
2. ST-elevation myocardial infarction (STEMI) within 30 days.
3. Planned treatment of additional lesions in the target vessel, or more than two (2) non-target lesions within non-target vessels, during the index procedure.
4. Target lesion is located within a bifurcation with planned treatment of side branch vessel.
5. Target lesion is the 3rd or greater stent failure (i.e., more than two [2] layers of stent are present at any segment of the target lesion).
6. Target vessel had any previous vascular brachytherapy treatment or is planned to undergo brachytherapy at index procedure.
7. Previous PCI of the target vessel within 30 days.
8. Planned PCI of a non-target vessel, or a non-target lesion in the target vessel, within 30 days of randomization.
9. Subject has chronic renal insufficiency (dialysis dependent, or glomerular filtration rate [GFR] ≤ 30 ml/min/1.73 m² within 30 days of index procedure) or has undergone renal transplantation.
10. Subject has acute renal insufficiency confirmed by 50% increase of serum creatinine within 48 hours before procedure and/or decrease in urine output.
11. History of active peptic ulcer or gastrointestinal bleeding within prior 6 months or other inability to comply with recommended duration of DAPT.
12. Subject is pregnant, breast-feeding, or a woman of childbearing potential who is not using appropriate contraceptives to avoid becoming pregnant.
13. Documented left ventricular ejection fraction (LVEF) < 25%.
14. Currently participating in another investigational drug or device study that has not completed primary endpoint follow-up.

Angiographic Exclusion Criteria

1. Target lesion is a total occlusion or has evidence of thrombus.
2. Target lesion involves an unprotected left main.
3. Target lesion has > 30% residual stenosis by visual estimate or dissection greater than NHLBI type C after pre-dilation/pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months post-index procedure

SECONDARY OUTCOMES:
Device success | Index Procedure
Lesion Success | Index Procedure
Procedure Success | Index Procedure
Composite Safety Endpoint | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
All-cause Mortality | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
Cardiovascular Mortality | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
MI | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
Clinically driven TLR, all TLR | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
Clinically driven TVR, all TVR, non-TVR | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
TLF | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
TVF | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
Stent Thrombosis | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
Bleeding | Prior to discharge, at 1, 6, and 12 months
Net adverse clinical events | Prior to discharge, at 1, 6, and 12 months and annually thereafter through 5 years follow-up
Binary angiographic restenosis | 12 months
In-stent percent diameter stenosis | 12 months
In-segment percent diameter stenosis | 12 months
In-stent LLL | 12 months
In-segment LLL | 12 months
In-stent MLD | 12 months
In-segment MLD | 12 months
OCT assessment of neointimal hyperplasia, neo-atherosclerosis, and stent malapposition | 12 months
TLF | 12 months
  SELUTION SLR 014 DEB versus DES among participants with one previous layer of stent

OTHER OUTCOMES:
Cardiac Biomarker Elevations | Peri-Procedural

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Cutlip, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (48):
- United States (34):
  - Loma Linda University, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California
  - ClinRe 001-001, Thornton, Colorado
  - MedStar Heart Institute, Washington D.C., District of Columbia
  - University of Florida Health, Jacksonville, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Ascension St Vincents Heart Center, Indianapolis, Indiana
  - Ascension Via Christi, Wichita, Kansas
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Centre, Harvard Medical School, Boston, Massachusetts
  - Ascension Borgess Heart Institute, Kalamazoo, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Ascension St John Hospital, Southfield, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Manchester Catholic Medical Center, Manchester, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Mount Sinai Hospital, New York, New York
  - St. Francis Hospital & Heart Center, Roslyn, New York
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Integris, Oklahoma City, Oklahoma
  - UPMC Pinnacle Health, Harrisburg, Pennsylvania
  - Pennsylvania State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lifespan Cardiovascular Institute, Providence, Rhode Island
  - HCA Centennial, Nashville, Tennessee
  - Baylor Scott & White, Dallas, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Baylor Scott & White, Temple, Texas
  - HCA Chippenham/VA Cardiovascular Specialists, Richmond, Virginia
- HartCentrum Hasslet, Jessa Ziekenhuis, Hasselt, Belgium
- Brazil (2):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto do Coração - São Paulo University, São Paulo, São Paulo
- Hamilton Health Sciences, Hamilton, Ontario, Canada
- France (4):
  - Clinique Valmy, Dijon
  - Hôpital privé Jacques Cartier, Massy
  - Clinique Saint Hilaire, Rouen
  - CHU Toulouse Rangueil, Toulouse
- Italy (3):
  - Maria Cecilia Hospital, Cotignola
  - Instituto Clinico Humanitas Milan, Milan
  - Center Azienda Ospedaliero Universitaria de Padova, Padua
- Netherlands (3):
  - Amsterdam UMC, Academic Medical Centre, Amsterdam, AZ
  - UMC Utrecht, Utrecht, CX
  - UMCG, Groningen, GZ

REFERENCES:
- [Derived] Cutlip DE, Mehran R, Doros G, Kaplinskiy V, Lee J, Zheng L, Kausik M, Osborn E, Waksman R. Prospective randomized single-blind multicenter study to assess the safety and effectiveness of the SELUTION SLR 014 drug eluting balloon in the treatment of subjects with in-stent restenosis: Rationale and design. Am Heart J. 2025 Jun;284:11-19. doi: 10.1016/j.ahj.2025.02.001. Epub 2025 Feb 12. PMID 39952378